CLINICAL TRIAL: NCT02118831
Title: Systemic Pharmacokinetics Following Intravitreal Injections of Ranibizumab, Bevacizumab or Aflibercept in Patients With Neovascular Age-related Macular Degeneration
Brief Title: Systemic Pharmacokinetics Following Intravitreal Injections of Anti-VEGF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ML28032
Record Dates: First submitted 2014-04-15; First posted 2014-04-21 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Age-related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
Keywords: macular degeneration; diabetic macular edema; vein occlusion; vascular endothelial growth factor
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion | interventions — aflibercept; Bevacizumab; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aflibercept Blood Sample Collection (Active Comparator): Blood samples will be collected from patients receiving aflibercept following the first and third dose of standard care therapy.
  Interventions: Biological: Blood Sample Collection; Drug: Aflibercept
- Bevacizumab Blood Sample Collection (Active Comparator): Blood samples will be collected from patients receiving bevacizumab following the first and third dose of standard care therapy.
  Interventions: Biological: Blood Sample Collection; Drug: Bevacizumab
- Ranibizumab Blood Sample Collection (Active Comparator): Blood samples will be collected from patients receiving ranibizumab following the first and third dose of standard care therapy.
  Interventions: Biological: Blood Sample Collection; Drug: Ranibizumab

INTERVENTIONS:
Biological: Blood Sample Collection — Subjects will have their blood drawn for analysis following their first and third injections of anti-VEGF.
Drug: Aflibercept — an intravitreal injection of Aflibercept administered three times on a monthly basis.
  Other Names: Eylea
  Arms: Aflibercept Blood Sample Collection
Drug: Bevacizumab — an intravitreal injection of Bevacizumab administered three times on a monthly basis.
  Other Names: Avastin
  Arms: Bevacizumab Blood Sample Collection
Drug: Ranibizumab — an intravitreal injection of Ranibizumab administered three times on a monthly basis.
  Other Names: Lucentis
  Arms: Ranibizumab Blood Sample Collection

SUMMARY:
Comparable data for bevacizumab and aflibercept are lacking, as are studies comparing the systemic levels of ranibizumab, bevacizumab, and aflibercept and their relative effects on circulating vascular endothelial growth factor. In the present prospective study, the investigators evaluated serum drug levels and plasma free vascular endothelial growth factor (VEGF) levels in patients with neovascular age-related macular degeneration following intravitreal injections of ranibizumab, bevacizumab and aflibercept.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent for participation in this study
* Subjects with a diagnosis of neovascular age-related macular degeneration, diabetic macular edema, or retinal vein occlusion who are either treatment naïve or more than 4 months out from a prior intravitreal anti-vascular endothelial growth factor injection

Exclusion Criteria:

* Subjects unwilling to receive 3 monthly injections of anti-vascular endothelial growth factor as initial therapy
* Subjects who may need or have received systemic anti-vascular endothelial growth factor for oncology in the past year
* Subjects with history of another ocular disease other than neovascular age-related macular degeneration, diabetic macular edema, or retinal vein occlusion
* Subjects with history of vitrectomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Avery, MD, Principal Investigator — California Retina Consultants; Melvin D Rabena, BS, Study Director — California Retina Consultants

REFERENCES:
- [Derived] Avery RL, Castellarin AA, Steinle NC, Dhoot DS, Pieramici DJ, See R, Couvillion S, Nasir MA, Rabena MD, Le K, Maia M, Visich JE. Systemic pharmacokinetics following intravitreal injections of ranibizumab, bevacizumab or aflibercept in patients with neovascular AMD. Br J Ophthalmol. 2014 Dec;98(12):1636-41. doi: 10.1136/bjophthalmol-2014-305252. Epub 2014 Jul 7. PMID 25001321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were recruited at a single private medical clinic between May of 2012 through October 2013
Groups:
- Aflibercept: Blood samples will be collected from patients receiving aflibercept following the first and third dose of standard care therapy.
  Aflibercept: Subjects will receive intravitreal aflibercept as part of their routine medical care.
- Bevacizumab: Blood samples will be collected from patients receiving bevacizumab following the first and third dose of standard care therapy.
  Bevacizumab: Subjects will receive intravitreal bevacizumab as part of their routine medical care.
- Ranibizumab: Blood samples will be collected from patients receiving ranibizumab following the first and third dose of standard care therapy.
  Ranibizumab: Subjects will receive intravitreal ranibizumab injections as part of their routine medical care.
Period: Overall Study
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Started | 21 | 15 | 20
Completed | 21 | 15 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab | Total
Number analyzed (Participants) | 21 | 15 | 20 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (4) | 75 (3) | 77 (5) | 76 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 10 | 27
  Male | 10 | 9 | 10 | 29
Region of Enrollment [Number; unit: participants]
  United States | 21 | 15 | 20 | 56

OUTCOME MEASURES:

1. Primary Outcome: Serum Pharmacokinetics Following Treatment From 1st and 3rd Doses
Description: Maximum serum levels of ranibizumab, bevacizumab or aflibercept will be measured after the first and third injections, up to 28 days following each treatment.
Time Frame: Up to 4 months
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 21 | 15 | 20
nM
  After 1st dose | 0.45 (0.29) | 0.76 (0.31) | 0.11 (0.13)
  After 3rd dose | 0.58 (0.52) | 1.47 (0.55) | 0.07 (0.05)

2. Secondary Outcome: Change in Minimum Serum Levels of Free Vascular Endothelial Growth Factor From Baseline to Month 4 (One Month After Last Treatment)
Description: Minimum serum levels of free vascular endothelial growth factor will be measured at baseline and at 4 months following treatment (one month after last treatment).
Time Frame: baseline and month 4
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Number analyzed (Participants) | 21 | 15 | 20
pg/mL
  Baseline | 19.2 [15.3 to 23.1] | 22.5 [17.3 to 27.6] | 17.0 [11.6 to 22.5]
  Month 4 | 11.3 [8.5 to 14.2] | 10.6 [6.9 to 14.1] | 17.0 [13.2 to 21.7]

ADVERSE EVENTS:
Arm/Group | Aflibercept | Bevacizumab | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/15 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/15 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes